CLINICAL TRIAL: NCT05943821
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Effect of Allopurinol on the Risk of Cardiovascular Events in Patients with High and Very High Cardiovascular Risk, Including the Presence of Long-COVID Syndrome.
Brief Title: The Effect of Allopurinol on the Risk of Cardiovascular Events in Patients with Cardiovascular Risk
Acronym: ALL-VASCOR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022/ABM/01/00027
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Cardiovascular Diseases; Uric Acid
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allopurinol (Active Comparator): The patients will receive allopurinol at an initial daily dose of 200 mg. If insufficient therapy efficacy is noted, the initial allopurinol dose will be increased by 100 mg (up to 300 mg during V2). Similarly, the dose may be increased by another 100 mg at visit 3 and by another 100 mg at the visit 4 (up to 500 mg during V4).
  Interventions: Drug: Allopurinol 200 mg; Drug: Optional intervention
- Placebo (Placebo Comparator): The patients will receive placebo at an initial daily dose of 200 mg. The dose may be increased by another 100 mg at visit 3 and by another 100 mg at the visit 4 (up to 500 mg during V4).
  Interventions: Drug: Allopurinol 200 mg; Drug: Optional intervention

INTERVENTIONS:
Drug: Allopurinol 200 mg — The intervention will occur after randomly allocating participants to the first group (G1), in which patients will receive allopurinol at an initial daily dose of 200 mg, or to the second group (G2), where they will receive a placebo. The placebo will be prepared as tablets with the same shape and appearance as the tested drug tablets, in the appropriate doses, and containing the same excipients. Participants will initially take one tablet of the medication daily in the morning. The physicians will dispense the drugs in packs of 30 tablets for the entire interval between visits (therapy 26 weeks ± 2 weeks). The patients will receive the medications during visit V1. The drugs will be prepared in identical packages, appropriately sealed, with a number for drug identification.
  Other Names: Allopurinol
Drug: Optional intervention — Approximately 26 weeks(+/-2 weeks) after the start of the intervention, the efficacy of the treatment will be evaluated at the follow-up visit V2. Efficacy is defined as achieving a serum UA level below 5.0mg/dL for those with baseline levels >5.0 to 7.0mg/dL or below 5.5mg/dL for those with baseline levels ≥7.0mg/dL. If insufficient therapy efficacy is noted, the initial allopurinol dose will be increased by 100mg (up to 300mg during V2). The dose may be increased by another 100mg at visit 3 and by another 100mg at the visit 4(up to 500mg during V4). In the placebo group, an appropriate preparation will be added so that the number of tablets corresponds to the group with the active substance.
  This treatment will be continued until the end of the bservation. Patients who meet their UA target concentration at visit V2 or V3, or V4, and those who fail to meet their target concentration at visit V4, will not have their dosing changed until the end of the follow-up.
  Other Names: Please describe in more detail

SUMMARY:
Numerous studies, but not all, have suggested a positive effect of allopurinol on the cardiovascular system. The ALL-VASCOR study aims to evaluate the efficacy of allopurinol therapy for improving cardiovascular outcomes in patients at high and very high cardiovascular risk, excluding ischemic heart disease. This is particularly important due to the high cost of cardiovascular disease treatment and its status as one of the leading causes of death.

DETAILED DESCRIPTION:
The ALL-VASCOR study is a randomized, double-blind, placebo-controlled, multi-center trial that examines the effect of allopurinol therapy (200-500mg of allopurinol daily) versus an equivalent dose of placebo on the risk of cardiovascular events in 1,116 patients aged 40-70, with serum uric acid levels above 5mg/dL and with high and very high risk for cardiovascular disease. The ALL-VASCOR study is further designed to assess the occurrence of long-COVID syndrome. The study is directed toward both primary and secondary as well as additional endpoints. Due to the duration of the study, the planned intervention will end on July 31,2028, unless the Safe Monitoring Board or other applicable authorities decide about it. Participant recruitment for the ALL-VASCOR study is set to begin in August of 2023 and will be conducted only within Poland.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 40-70 years old.
2. Giving informed consent to participate in the study.
3. Serum UA levels above 5 mg/dl within the last six months before the screening visit.
4. Meeting at least one of the criteria defining high or very high CV risk includes:

   1. calculated 10-year cardiovascular mortality risk based on SCORE2 >2.5% for patients under 50 years old or ≥5% for patients 50 years old or older
   2. documented occurrence of CV diseases (cerebrovascular disease: ischemic stroke, intracerebral bleeding, TIA; heart failure regardless of the etiology NYHA I - II (without IHD), PAD, atrial fibrillation (de novo or ever)
   3. diabetes or arterial hypertension complicated by organ damage:

      * increase in vascular stiffness: pulse pressure ≥ 60 mmHg, and/or cervicofemoral PWV > 10 m/s;
      * features of left ventricular hypertrophy on echocardiography or electrocardiography;
      * increased urine albumin-creatinine ratio (30-300 mg/g);
      * ankle-brachial index < 0.9.

Exclusion Criteria:

1. Taking allopurinol, febuxostat or other hypouricemic drugs.
2. Contraindications to taking allopurinol.
3. Pregnant women, breastfeeding or planning pregnancy during the duration of the study.
4. Hormonal therapy containing oestrogens.
5. Active cancer process or disease in the last five years, excluding locally malignant tumours.
6. Uncontrolled hypertension (mean value ≥ 180/110 mmHg seven days before screening visit) in home measurements despite using hypotensive drugs.
7. 7. Renal insufficiency with an eGFR <45 ml/ min/1.73m2 (according to 2009 CKD-EPI recommendations: stage G3b, G4 and G5).
8. Hypothyroidism or hyperthyroidism not in a state of euthyroidism.
9. Confirmed coronary artery disease (defined as prior AMI, revascularization of the myocardium, confirmed presence of atherosclerotic plaques in coronary arteries on imaging studies).
10. Heart failure in NYHA class III and IV.
11. Taking preparations: azathioprine, mercaptopurine or cyclosporin. Participation in another clinical trial of a medicinal product or medical device within the last three months or five half-lives, whichever period is longer.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of a major adverse cardiovascular event (MACE) | Baseline up to approximately 5 years
  The number of all causes of death, cardiac death, stroke, transient ischemic attack, acute coronary syndrome, coronary angioplasty or revascularization, peripheral arterial angioplasty, hospitalization for unstable angina or worsening heart failure

SECONDARY OUTCOMES:
Percentage of Participants of all-cause death | Baseline up to approximately 5 years
  Events were adjudicated by researchers as all-cause death. The number of all-cause deaths recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11.
Percentage of Participants With Cardiac Death | Baseline up to approximately 5 years
  Description:Events were adjudicated by researchers as cardiac death. The number of all-cause deaths recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11.
Percentage of Participants With stroke | Baseline up to approximately 5 years
  Description:Events were adjudicated by researchers as stroke. The number of all-stroke recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11
Percentage of Participants With transient ischemic attack | Baseline up to approximately 5 years
  Description:Events were adjudicated by researchers as transient ischemic attack. The number of transient ischemic attack recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11
Percentage of Participants With acute coronary syndrome | Baseline up to approximately 5 years
  Description:Events were adjudicated by researchers as acute coronary syndrome,. The number of acute coronary syndrome, recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11
Percentage of Participants With coronary angioplasty or revascularization | Baseline up to approximately 5 years
  Description:Events were adjudicated by researchers as coronary angioplasty or revascularization. The number of coronary angioplasty or revascularization, recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11
Percentage of Participants With peripheral arterial angioplasty | Baseline up to approximately 5 years
  Description:Events were adjudicated by researchers as peripheral arterial angioplasty. The number of peripheral arterial angioplasty recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11
Percentage of Participants With hospitalization for unstable angina or worsening heart failure | Baseline up to approximately 5 years
  Events were adjudicated by researchers as endpoint hospitalization (hospitalization and stay in the emergency department due to heart failure, need for intravenous loop diuretics and/or doubling the dose of oral loop diuretics).
  The number of hospitalization for unstable angina or worsening heart failure recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11
Percentage of Participants With Hospitalization | Baseline up to approximately 5 years
  Events were adjudicated by researchers as endpoint hospitalization. The number of hospitalization for reasons other than the endpoint number 9, recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11

OTHER OUTCOMES:
Assessment of progression and/or development of organ complications and atherosclerosis, including: echocardiography | Baseline up to the follow-up visit number 7 - approximately 3 years
  assessment of echocardiographic parameters - analysis of changes in echocardiographic parameters assessed in transthoracic echocardiographic examination (TTE).Assessment of systolic function (ejection fraction) and left ventricular hypertrophy. Analysis of changes from the baseline
Assessment of progression and/or development of organ complications and atherosclerosis, including the assessment of incidence of atrial fibrillation | Baseline up to the follow-up visit number 7 - approximately 3 years
  the assessment of the incidence of atrial fibrillation in an electrocardiographic examination (documented incident of de novo atrial fibrillation during observation)
Assessment of progression and/or development of organ complications and atherosclerosis, including the assessment of end-stage kidney disease | Baseline up to the follow-up visit number 7 - approximately 3 years
  the assessment of end-stage kidney disease based on eGFR measurements. Analysis of changes from the baseline
Assessment of progression and/or development of organ complications and atherosclerosis, including Ultrasound examination | Baseline up to the follow-up visit number 7 - approximately 3 years
  The assessment of abdominal aorta diameter. Analysis of changes from the baseline
Assessment of progression and/or development of organ complications and atherosclerosis, including Doppler ultrasound of carotid arteries | Baseline up to the follow-up visit number 7 - approximately 3 years
  Assessment of intima-media complex and atherosclerotic plaques. Analysis of changes from the baseline
Assessment of progression and/or development of organ complications and atherosclerosis, including the assessment of ankle-brachial index | Baseline up to the follow-up visit number 7 - approximately 3 years
  Assessment of ankle-brachial index. Analysis of changes from the baseline
Assessment of progression and/or development of organ complications and atherosclerosis, including the assessment of pulse wave velocity | Baseline up to the follow-up visit number 7 - approximately 3 years
  the assessment of pulse wave velocity. Analysis of changes from the baseline
Occurrence of long-COVID symptoms | Baseline up to approximately 5 years
  Occurrence of long-COVID symptoms assessed based on a survey. Analysis of changes from the baseline. The survey will be recorded from visit 0 (screening visit) to the last follow-up visit. Depending on the patient and the time of enrollment into the study, this corresponds to visit 7-11
The assessment of treatment efficacy | Baseline up to the follow-up visit number 7- approximately 3 years
  Attainment of target serum UA levels of 5 mg/dL or 5.5 mg/dL, depending on baseline values
Assessment of the laboratory parameters | Baseline up to the follow-up visit number 7 - approximately 3 years
  Assesment of:
  Estimated glomerular filtration rate (eGFR). Albumin to creatinine ratio and urinary albuminuria. Glycosylated hemoglobin (HbA1c). Lipid profile. Plasma C-reactive protein concentrations. Activity of aspartate and alanine transaminases (AST, ALT) Analysis all parameters of changes from the baseline
Assessment of frequency of side effects | From the first dose of allopurinol or placebo until the end of the observation period (approximately 3-5 years)
  Proportion of subjects who experienced at least one serious adverse event (SAE) during the study
Assessment of changes in participants' cardiovascular risk | Baseline up to approximately 5 years
  Assessment of changes in participants' cardiovascular risk based on the SCORE 2 scale. Analysis of changes from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Tykarski, Prof MD, Study Director — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewandowska K, Lipski D, Uruski P, Narkiewicz K, Januszewicz A, Wolf J, Prejbisz A, Rajzer M, Wiecek A, Tykarski A. Randomised, double-blind, placebo-controlled study evaluating the effect of allopurinol on the risk of cardiovascular events in patients with high and very high cardiovascular risk, including the presence of long-COVID-19 syndrome: the ALL-VASCOR study protocol. BMJ Open. 2024 Jul 24;14(7):e075741. doi: 10.1136/bmjopen-2023-075741. PMID 39053954